CLINICAL TRIAL: NCT04952844
Title: Functional Capacity in Survivors of COVID-19 Related ARDS: A Cross-sectional Study
Brief Title: Functional Capacity in Survivors of COVID-19 Related ARDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.014.IRB1.008
Record Dates: First submitted 2021-07-03; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Functional Capacity; Post-intensive Care Syndrome
Keywords: COVID-19; Acute Respiratory Distress Syndrome; 6-minute walk test; handgrip strength; MRC sumscore
MeSH Terms: conditions — COVID-19; postintensive care syndrome; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Acute respiratory distress syndrome survivors frequently develop impaired physical function, muscle weakness and quality of life. The aim of this retrospective study is to determine the functional capacity, global muscle weakness and quality of life of COVID-19 survivors after 4 weeks following hospital discharge and the relationship between different tools. COVID-19 related acute respiratory distress syndrome survivors were assessed 4 weeks following discharge from the hospital, 15 patients who attended the evaluation will be included the study. All subjects underwent standardized physical clinical evaluation, Medical Research Council-sumscore, hand-grip strength, 6-minute walk test, chair-stand test, timed up and go test and Short form-36, 4 weeks after hospital discharge.

DETAILED DESCRIPTION:
COVID-19 could cause acute respiratory distress syndrome in a minority of patients. After recovery from acute critical illness and discharged from hospital, secondary disabilities related to Post Intensive Care Syndrome could take over the role. There is limited data and information about the functional capacity of these patients after hospital discharge.Follow-up these patients after discharge might help assessing the symptoms of Post Intensive Care Syndrome, functional capacity and need of physical therapy, therefore give care for the impairments. The aim of this retrospective cross-sectional study is to demonstrate the functional capacity, global muscle weakness and quality of life of COVID-19 survivors after 4 weeks following hospital discharge and the relationship between different tools. Appointment was given all of the ARDS survivors related to COVID-19 who treated in ICU after 4 weeks following discharge from hospital in order to assess the need of rehabilitation. 15 patients who attended the evaluation will be included the study.

ELIGIBILITY:
Inclusion Criteria:

* to be older that 18 years
* Acute respiratory distress syndrome survivors related to COVID-19 who treated in Intensive care unit and attend appointment after 4 weeks following discharge from hospital

Exclusion Criteria:

* History of diseases that could affect functional capacity, muscle strength and quality of life, such as cancer, spinal cord disease, neuromuscular diseases
* do not want to attend the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute respiratory distress syndrome survivors related to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | 1 day
  Six-minute walk test is a field test evaluating submaximal aerobic capacity. The technical standards are defined by European Respiratory Society and American Thoracic Society. The individuals were asked to walk as far as possible in a 30-meter corridor in 6 minutes and the distance, oxygen saturation, heart rate, systolic blood pressure and dyspnea scale (Borg 0-20) were recorded before and immediately after the test, and recovery period (1. minute of recovery). It is a valid and responsive measurement of functional capacity and also predicts quality of life in Acute respiratory distress syndrome survivors

SECONDARY OUTCOMES:
Handgrip strength | 1 day
  Handgrip strength will be measured using a handheld dynamometer according to the instructions of the American Society of Hand Therapists. Patients will be requested to seat placing their arms by their sides with the elbow flexed to 90°, the forearm mid-prone, and the wrist in neutral position. Using standard verbal encouragement, patients will be asked to grip the dynamometer with dominant hand with maximal effort. Three trials will be performed with a 30-second interval between trials and the highest value will be recorded in kg. The cut-off values of grip strength are 28.6 kg in men and 16.4 kg in women.
Medical Research Council-sumscore | 1 day
  It is valid and reliable tool in survivors of critical illness, it will be used in order to evaluate the overall muscle strength
Short form - 36 | 1 day
  Short form - 36 measures health related quality of life. It is a self-reported survey that evaluates individual health status with eight parameters consisting of physical function, pain, role limitations attributed to physical problems, role limitations attributed to emotional problems, mental health, social functioning, energy/ vitality, general health perception. There is not a summary score, each section is scored between 0-100, 0 indicates the worst condition, 100 indicates the best.
Chair stand test | 1 day
  It is used to evaluate strength and endurance of lower limbs. Patients will be asked to sit on a chair with a 46 cm seat height by crossing their hands over their chest and stand and sit five times consecutively as fast as possible. The test starts in the sitting position and terminate at the last sitting position and the time will be recorded.
timed up and go test | 1 day
  The test will be used to assess physical function. It is an objective, reliable and simple test to evaluate both balance and functional movement. The patients will be asked to get up from a chair, walk 3 m, turn around, walk back and sit on the chair again. The time will be recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Held N, Moss M. Optimizing Post-Intensive Care Unit Rehabilitation. Turk Thorac J. 2019 Apr 1;20(2):147-152. doi: 10.5152/TurkThoracJ.2018.18172. Print 2019 Apr. PMID 30958989
- [Background] Ngai JC, Ko FW, Ng SS, To KW, Tong M, Hui DS. The long-term impact of severe acute respiratory syndrome on pulmonary function, exercise capacity and health status. Respirology. 2010 Apr;15(3):543-50. doi: 10.1111/j.1440-1843.2010.01720.x. Epub 2010 Mar 19. PMID 20337995
- [Background] Turan Z, Topaloglu M, Ozyemisci Taskiran O. Medical Research Council-sumscore: a tool for evaluating muscle weakness in patients with post-intensive care syndrome. Crit Care. 2020 Sep 18;24(1):562. doi: 10.1186/s13054-020-03282-x. No abstract available. PMID 32948221
- [Background] Wilcox ME, Herridge MS. Lung function and quality of life in survivors of the acute respiratory distress syndrome (ARDS). Presse Med. 2011 Dec;40(12 Pt 2):e595-603. doi: 10.1016/j.lpm.2011.04.024. Epub 2011 Nov 9. PMID 22078086
- [Background] Chan KS, Zheng JP, Mok YW, Li YM, Liu YN, Chu CM, Ip MS. SARS: prognosis, outcome and sequelae. Respirology. 2003 Nov;8 Suppl(Suppl 1):S36-40. doi: 10.1046/j.1440-1843.2003.00522.x. PMID 15018132
- [Background] Hui DS, Wong KT, Ko FW, Tam LS, Chan DP, Woo J, Sung JJ. The 1-year impact of severe acute respiratory syndrome on pulmonary function, exercise capacity, and quality of life in a cohort of survivors. Chest. 2005 Oct;128(4):2247-61. doi: 10.1378/chest.128.4.2247. PMID 16236881